CLINICAL TRIAL: NCT00179842
Title: Immune Ablation and Hematopoietic Stem Cell Support in Patients With Severe Crohn's Disease
Brief Title: Immune Ablation and Stem Cell Support for Crohn's Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BMT 1202
Record Dates: First submitted 2005-09-10; First posted 2005-09-16 (Estimated); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Stem Cell Transplant

SUMMARY:
The investigators anticipate that this study will also form the basis to clarify further the role of the immune system in Crohn's disease.

DETAILED DESCRIPTION:
This study is designed to ablate an aberrant immune system and then, similar to the use of marrow transplants for immunodeficient patients, reconstitute a new immune system with lymphocyte depleted stem cells. Subsequent disease activity will be followed by (1) Crohn's disease activity index (CDAI), (2) quality of life instrument (IBDQ), (3) type and amount of therapy for CD, and (4) flow cytometry of peripheral blood lymphocyte subsets. In addition, the subjects will undergo periodic absorption function testing, to assess small intestinal function. We anticipate that this study will also form the basis to clarify further the role of the immune system in Crohn's disease.

ELIGIBILITY:
Inclusion Criteria:

* Less than physiologic age 60 at time of pretransplant evaluation.
* An established clinical diagnosis of severe CD that has failed therapy with prednisone, azathioprine, 5 ASA products and metronidazole, and has failed to have a sustained decrement of 70 points in the CDAI after one course of anti-TNF alpha, Infliximad. The patient is being considered for therapy with cyclosporin A (CSA) or surgical resection. The CDAI (appendix A) is 250-400.
* Pre-study peripheral blood counts must include a platelet count greater than 100,000/ul and an absolute neutrophil count greater than 1500/ul.
* Stem cell harvest greater than 1.4 x 106 CD34 cells/kg after CD34+ selection (to continue to transplant.)

Exclusion Criteria:

* HIV positive
* History of coronary artery disease, or congestive heart failure.
* Uncontrolled diabetes mellitus, or any other illness that in the opinion of the investigators would jeopardize the ability of the patient to tolerate aggressive chemotherapy
* Prior history of malignancy except localized basal cell or squamous skin cancer. Other malignancies for which the patient is judged to be cured by local surgical therapy, such as head and neck cancer, or stage I breast cancer will be considered on an individual basis.
* Positive pregnancy test, lactation, inability or unwillingness to pursue effective means of birth control, failure to accept or comprehend irreversible sterility as a side effect of therapy.
* Psychiatric illness or mental deficiency making compliance with treatment or informed consent impossible.
* FEV I/FVC < 50% of predicted, DLCO < 50% of predicted.
* Resting LVEF < 40%
* Bilirubin > 2.0 mg/dl, transferase (AST) > 2x upper limit of normal, unless the abnormalities are secondary to Crohn's disease.
* Serum creatinine > 2.0 mg/dl.
* Platelet count less than 100,000/ul, ANC less than 1500/ul.
* Patients presenting with intestinal perforation or toxic megacolon, or a suppurative problem that will require urgent surgery. In addition, the patient may not have any active infection. The presence of intestinal stomas does not exclude the patient from study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2007-03-22 (Actual); Primary Completion 2008-12-19 (Actual); Study Completion 2008-12-19 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and efficacy of treating severe CD with high dose cyclophosphamide and antithymocyte globulin rescued with T cell depleted autologous stem cells. Data will be used to evaluate the efficiency of a future phase III protocol. | Minimum of 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Sonali Chaudry, M.D., Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H Lurie Children's Hospital of Chicago, Chicago, Illinois, United States